CLINICAL TRIAL: NCT00758888
Title: Effect of Orthopedic Blocking on Cervical Spine Flexion and Extension Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Kristan Giggey, DC, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD0801080145
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2008-09

CONDITIONS: Sacroiliac Function

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment (Experimental): Place the blocks under the pelvis for 2 minutes
  Interventions: Procedure: Orthopedic Blocking
- Trochanter Belt (Active Comparator): Participant is fitted with trochanter belt on the adjusting table and wear it while Investigator checks their flexion and extension strength.
  Interventions: Procedure: Trochanter Belt
- Sham (Sham Comparator): Participant lies on adjusting table, blocks are placed in a similar configuration but distant to actual points of leverage.
  Interventions: Other: Blocking Sham

INTERVENTIONS:
Procedure: Orthopedic Blocking — Place the blocks under the pelvis for 2 minutes
  Arms: Treatment
Procedure: Trochanter Belt — Participant is fitted with trochanter belt on the adjusting table and wear it while Investigator checks their flexion and extension strength.
  Arms: Trochanter Belt
Other: Blocking Sham — Participant lies on adjusting table, blocks are placed in a similar configuration but distant to actual points of leverage.
  Arms: Sham

SUMMARY:
A few studies concerning the effects of joint manipulation have shown muscle responses distal to the site of manipulation. The purpose of this study is to determine if pelvic orthopedic blocking, a low force method of manipulating the sacroiliac joint, can have produce changes to cervical spine function.

DETAILED DESCRIPTION:
All mechanoreceptor types are found in diarthrodial joints. Mechanoreceptor afferents have reflexive connections to motor neurons. Stimulation of muscle and joint afferents are known to produce reflexive muscle changes. Orthopedic blocking applies a gentle compression to the sacroiliac joints. The current study seeks to determine if orthopedic blocking of the sacroiliac joint can affect cervical spine function thereby serving as a useful adjunctive procedure in the treatment of cervical spine joint dysfunction. The current study will compare pre & post treatment cervical isometric strength readings from an orthopedic blocking group, a trochanter belt group (another type of compression), and a sham group.

ELIGIBILITY:
Inclusion Criteria:

* Logan faculty, students, or staff 18-30 years of age with a leg-length inequality of 5mm or more.

Exclusion Criteria:

* Fractures
* Tumors
* Myopathies
* Consumption of prescription drugs that affect nervous system function
* Recent cervical spine injuries or surgeries
* Cervical pain

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Cervical Isometric Strength | Pre and post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States